CLINICAL TRIAL: NCT05795634
Title: Cognitive Vulnerability to Stress in Individuals at Risk for Alzheimer's Disease (Stress-AD)
Brief Title: Cognitive Vulnerability to Stress in Individuals at Risk for Alzheimer's Disease
Acronym: Stress-AD
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Johns Hopkins University (Other)
Collaborators: National Institute on Aging (NIA) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: IRB00313479; R01AG065171 (NIH)
Record Dates: First submitted 2023-03-07; First posted 2023-04-03 (Actual); Last update posted 2026-01-29 (Actual); Status verified 2026-01

CONDITIONS: Mild Cognitive Impairment; Alzheimer Disease
Keywords: Stress; Neuropsychology; Endocrine; Genetics; Blood biomarkers
MeSH Terms: conditions — Cognitive Dysfunction; Alzheimer Disease | interventions — Psychological Tests

STUDY DESIGN:
Intervention Model Description: Prospective study using baseline characteristics to predict outcomes
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Trier Social Stress Test (Other): All participants in the study will get undergo the same stress procedure
  Interventions: Behavioral: Trier Social Stress Test

INTERVENTIONS:
Behavioral: Trier Social Stress Test — Acute psychosocial stress procedure; 5 minutes of public speaking and 5 minutes of mental arithmetic

SUMMARY:
The goal of this clinical trial is to learn about how genetics and the response to stress predicts cognitive decline in individuals with mild cognitive impairment.

The main question[s] it aims to answer are:

* Does the hormone response to acute stress predict the degree of cognitive impairment following acute stress?
* Do genes associated with the risk for Alzheimer's disease influence the relationship between stress hormone response to stress and cognitive impairment following stress?
* Do cognitive impairment following acute stress and genes associated with the risk for Alzheimer's disease predict cognitive decline and change in biomarkers for Alzheimer's disease 2 years later?

Participants will have 3 in-person study visits. The first 2 will occur at baseline and the 3rd visit will occur 2 years later. During the visits, participants will provide blood and saliva samples, undergo a 10-minute social stress procedure, complete questionnaires, and take tests of memory and other thinking skills. Someone who knows the participant (a "study partner") will be asked questions about the participant's daily functioning at the first and 3rd study visits.

DETAILED DESCRIPTION:
In the wake of discouraging results from treatment trials in Alzheimer's disease (AD), there is emerging consensus that the lack of efficacy in these trials is attributable to heterogeneity in the course of AD. Among the potential causes of heterogeneity, the investigators aim to focus on vulnerability to acute stress. Although associations between stress and the risk of AD are well established, these findings have not been used to inform AD intervention efforts. The investigators aim to address this crucial gap. Considering that in healthy individuals, acute stress can impair cognition in those who have risk factors for AD, the investigators propose that these individuals may represent a specific endophenotype who could be targeted for AD treatment trials. The investigators' prior findings implicate the endocrine stress response as an important component of AD risk that warrants further study.

The investigators aim to conduct a prospective study to examine the associations among the acute endocrine stress response, cognitive impairment following acute stress, and subsequent cognitive decline. For the investigators' basic study design, the investigators will induce acute stress with the Trier Social Stress Test (TSST; 5 minutes of public speaking and 5 minutes of mental arithmetic) and then administer a battery of cognitive tests. Two cognitive domains-memory and executive functioning-will be the primary cognitive outcomes. Salivary samples collected at fixed intervals will be used to measure stress hormone response; cortisol will the primary endocrine hormone outcome. The investigators will also examine the influence of apolipoprotein E (APOE) gene polymorphisms and polygenic risk scores, conduct sex-stratified analyses, and collect blood-based biomarkers for AD.

The investigators' study has 3 primary aims:

1. To determine the association between endocrine response to acute stress and memory and executive test performance following acute stress in individuals with MCI due to AD.
2. To examine the moderating effect of APOE genotype and polygenic risk score derived from genome wide genotyping on the association between endocrine response to acute stress and cognitive test performance following acute stress in individuals with MCI due to AD.
3. To determine predictors of cognitive decline and neurodegeneration at 2-year follow-up.

Secondary Aims: Conduct the analyses from Specific Aims 1-3 in men and women separately in order to identify sex-specific predictors of stress-induced memory and executive impairment and cognitive decline after 2 years. As an exploratory aim, the investigators will examine the influence of personality factors and stressful life events on the hypothesized associations.

For this study, participants will come to the clinic for 3 study visits. For the first visit, participants will be asked to bring someone who knows the participant well (a "study partner"). During that visit, participants and the participants' study partners will answer questions about the participant's daily functioning. In addition, participants (but not the participants study partners) will take paper-and-pencil tests and provide a blood sample. About one month later, participants will return for a second study visit, but the participants' study partner does not need to come to that visit. During that second visit, participants will undergo a brief procedure (public speaking and mental math) that is designed to cause stress, during which the investigators will measure participants' stress hormones by asking participants to provide the investigators with samples of the participants' saliva. Two years later, participants and the participants' study partners will return for Visit 3. At that visit, the investigators will ask participants to provide another blood sample and complete tests of memory and other thinking skills. Study partners will answer questions about the participants during this visit but will not take any tests or provide a blood sample.

ELIGIBILITY:
Inclusion Criteria for Subjects with Mild Cognitive Impairment (MCI)

* Age 60 and older
* Fluent English speaker
* Able to provide informed consent for study procedures
* Willing and able to return for 2-year-followup visit
* Willing and able to provide an informant who can participate in the screening and 2-year study visits
* BMI >17 and <30
* Meets clinical and cognitive criteria for mild cognitive impairment (MCI) using National Institute on Aging (NIA)/Alzheimer's Association 2011 criteria (see below)

Exclusion Criteria for Subjects with MCI

* Current smoker
* Current or past history of major psychiatric illness, including schizophrenia, bipolar disorder, obsessive-compulsive disorder, post-traumatic stress disorder
* Neurological disorder, including Parkinson's disease, Huntington's disease
* Current or past history of immune disorder, including multiple sclerosis
* Current or past history of drug dependence
* Treatment within the last six months with: neuroleptics, sedative hypnotics, or glucocorticoids
* History of head injury with loss of consciousness for more than ½ hour, stroke, or seizure
* General surgery within the last 3 months
* Sensory impairment (poor vision or hearing) significant enough to interfere with ability to provide valid cognitive test data

Clinical and Cognitive Criteria for MCI due to AD

* Cognitive concern reflecting a change in cognition reported by patient or informant or clinician (i.e., historical or observed evidence of decline over time)
* Objective evidence of impairment in one or more cognitive domains, typically including memory (i.e., formal or bedside testing to establish level of cognitive function in multiple domains)
* Preservation of independence in functional abilities
* Not demented
* Etiology of MCI consistent with AD pathophysiological process

Inclusion Criteria for Study Partners

* Age 21 or older
* Able to participate in an interview
* Willing and able to attend study visits
* Willing and able to return for 2-year-followup visit

Exclusion Criteria for Study Partners

• Unwilling to answer questions about the participant with MCI

Min Age: 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 240 (Estimated)
Dates: Start 2023-03-01 (Actual); Primary Completion 2028-03-01 (Estimated); Study Completion 2029-03-01 (Estimated)

PRIMARY OUTCOMES:
Change in mean memory test composite score | Baseline and Visit 2 (up to 1 month) and Baseline to Visit 3 (up to 2 years)
  Change in the mean composite score of the following memory tests: Neuropsychological Assessment Battery Word List Memory test, Morris Revision test, and a computerized Pattern Separation Task, with higher composite score indicating better memory
Change in mean executive test composite score | Baseline and Visit 2 (up to 1 month) and Baseline to Visit 3 (up to 2 years)
  Change in the mean composite score of the following executive tests: phonemic (letter) fluency test, part B of the Trial Making Test, and the backwards trial of a Digit Span task, with higher composite score indicating better executive functioning

SECONDARY OUTCOMES:
Change (in nanogram per liter; ng/L) in level of neurofilament light (NF-L) | Baseline to Visit 3 (up to 2 years)
  Change in a blood biomarker of neurodegeneration, with higher levels indicating greater neurodegeneration

CONTACTS AND LOCATIONS:
Overall Officials: Cynthia A Munro, PhD, Principal Investigator — Johns Hopkins School of Medicine
Locations (1):
- Johns Hopkins School of Medicine, Baltimore, Maryland, United States

IPD SHARING:
Plan to Share IPD: Yes
Study investigators are committed to resource sharing, according to NIH policy. At the conclusion of the study, after the final freeze to the database, a public use database will be created and made available along with specifications for its use. Johns Hopkins University will share anonymized genomic sequence data by depositing these data in the database of Genotypes and Phenotypes (dbGaP) (a controlled-access database funded by NIH).
  In addition, the investigators will share data from biosamples (saliva and blood samples), including genotype data, at the time of publication of the primary results or within 9 months of database lock, whichever comes first. These data will be shared via the Alzheimer's Clinical Trials Consortium (ACTC), and/or the National Alzheimer's Coordinating Center (NACC).
Supporting Information: Study Protocol
Time Frame: At time of publication of primary results or within 9 months of database lock, whichever comes first. No end data for data availability has been determined at this time.
Access Criteria: Researchers at academic institutions are eligible.